CLINICAL TRIAL: NCT04399577
Title: Complement Component 3c and Tumor Necrosis Factor-α in Patients With Human Papillomavirus-Induced Cutaneous Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha M Hammad, MD, Principal investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3140/23-10-2016
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — PRA1 protein, Candida albicans

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wart Patients (Experimental): Patient receive 0.1 mL of diluted preparation of candida solution at 2 weeks interval for the maximum of 5 sessions
  Interventions: Biological: Candida antigen

INTERVENTIONS:
Biological: Candida antigen — Patient receive candida antigen immunotherapy and blood samples will be withdrawn before and after intervention

SUMMARY:
The investigators explore the role of the complement pathway and T helper 1 immune response in clinical response to Candida immunotherapy via complement component and tumor necrosis factor, respectively.

DETAILED DESCRIPTION:
39 patients are enrolled in the study They suffer from chronic recurrent cutaneous warts Patients receive Candida antigen immunotherapy vial intra-lesional injection every 2 weeks till complete resolution or the maximum of 5 sessions Blood samples are withdrawn before and after intervention C3, C4, MBL, C3C and TNF alpha serum levels are measured

ELIGIBILITY:
Inclusion Criteria:

* Chronic multiple cutaneous

Exclusion Criteria:

* Hypersensitivity to Candida antigen
* Fever
* Immunosuppressive disorders
* Previous wart therapy in the last month

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Resolution of warts | 12 weeks
  100% clearance of warts

SECONDARY OUTCOMES:
Recurrence | 6 months
  Reappearance of warts

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Derived] Hammad NM, Abdelhadi AA, Fawzy MM, Marei A. Complement component 3c and tumor necrosis factor-alpha systemic assessment after Candida antigen immunotherapy in cutaneous warts. Braz J Microbiol. 2020 Dec;51(4):1673-1681. doi: 10.1007/s42770-020-00322-0. Epub 2020 Jun 27. PMID 32594377